CLINICAL TRIAL: NCT07032376
Title: Guideline to Implementation: A Rapid Clinical Care Pathway to Care for Patients Affected by Chronic Constipation- Phase 2
Brief Title: A Rapid Clinical Care Pathway to Care for Patients Affected by Chronic Constipation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Eric Shah, Associate Professor of Internal Medicine, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00228948b; 1K23DK134752-01 (NIH)
Record Dates: First submitted 2025-06-19; First posted 2025-06-24 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Constipation
Keywords: Questionnaires; Gastroenterology care; Rectal Expulsion Device (RED)
MeSH Terms: conditions — Constipation | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chronic constipation (Experimental): Participants will complete surveys and may or may not have the Rectal Expulsion Device (FDA 510k approved) used during clinic visit.
  Interventions: Behavioral: Survey; Behavioral: Rectal Expulsion Device use

INTERVENTIONS:
Behavioral: Survey — All participants will complete a baseline survey and have medical information collected.
Behavioral: Rectal Expulsion Device use — During the participant's clinic visit for constipation, the Rectal Expulsion Device will be available for the gastroenterology care provider to use if the decision is made to use this during the clinic visit.
  In addition, the care provider will have access to the RED brochure and the Michigan Chart (MICHART) Our Practice Advisory (OPA) - a decision support tool in MiChart to support care navigation using RED.

SUMMARY:
This research is studying how the availability of a Food and Drug Administration (FDA)-cleared point-of-care, bedside device bedside device called Rectal Expulsion Device (RED) can be used to evaluate constipation in the participants' routine office visit with the participants' care provider. In this research, participants will be asked to complete a survey prior to the gastroenterology office consultation. Health-related information will be collected for this research study. There are no additional study visits for this research study.

DETAILED DESCRIPTION:
This registration is (Implementation Phase) for the registered study "Guideline to Implementation: A Rapid Clinical Care Pathway to Care for Patients Affected by Chronic Constipation" (Observational Phase) NCT06352827.

ELIGIBILITY:
Inclusion Criteria:

* Participant has Chronic constipation as a main symptom
* Participant is able to participate in pelvic floor physical therapy

Exclusion Criteria:

* Participant has taken narcotic pain medication in the past 30 days
* Participant has been scheduled for a test called an anorectal manometry in the past
* Participant has been scheduled to see a pelvic floor physical therapist in the past
* Participant is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of encounters in which anorectal physiology testing is ordered or performed at the baseline routine-care gastroenterology office appointment | Day 1 (Baseline = initial appointment after consent)]
  Fidelity to ordering pelvic floor diagnostics
Percentage of encounters in which pelvic floor physical therapy is ordered at the baseline routine-care gastroenterology office appointment | Day 1 (Baseline = initial appointment after consent)]
  Fidelity to ordering pelvic floor treatment

CONTACTS AND LOCATIONS:
Overall Officials: Eric Shah, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No